CLINICAL TRIAL: NCT07075185
Title: A Phase 1 Study to Evaluate the Safety of KLN-1010, a Novel, In Vivo Gene Therapy to Generate Anti-B Cell Maturation Antigen (Anti-BCMA) Chimeric Antigen Receptor-T Cells (CAR-T) in Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: A Study to Evaluate a Novel Gene Therapy in Patients With Relapsed and Refractory Multiple Myeloma
Acronym: inMMyCAR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kelonia Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KLN-001
Record Dates: First submitted 2025-07-02; First posted 2025-07-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma in Relapse; Myeloma Multiple; Multiple Myeloma Progression; Neoplasms by Histologic Type; Neoplasm; Hemostatic Disorders; Vascular Disorder; Paraproteinemias; Blood Protein Disorders; Hematologic Disease and Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Disease; Gene Therapy
Keywords: in vivo CAR-T; multiple myeloma; gene therapy; BMCA
MeSH Terms: conditions — Multiple Myeloma; Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorders; Vascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Disease; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- KLN-1010 (Experimental): Drug: KLN-1010 specified dose given once
  Interventions: Drug: KLN-1010

INTERVENTIONS:
Drug: KLN-1010 — Given at specified dose one time

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and recommended Phase 2 Dose (RP2D) of KLN-1010 in patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have relapsed and refractory multiple myeloma (RRMM) with measurable disease
* Participants must have received at least 3 prior lines of therapy including a proteasome inhibitor (PI), an immunomodulatory drug (IMiD), and CD38-directed monoclonal antibody
* Participants must have an Eastern Cooperative Group (ECOG) performance status of 0-1
* Participants must have acceptable laboratory values as defined by the protocol

Exclusion Criteria:

* Participants must not have known central nervous system (CNS) involvement with myeloma
* Participants cannot have plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, and skin changes) syndrome, or primary light chain amyloidosis
* Participants cannot have ongoing acute systemic infection requiring antimicrobial therapy
* Participants cannot require systemic steroids for any condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2042-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs), including dose-limiting toxicities (DLTs), and/or establish the recommended Phase 2 Dose | Up to 15 years from dosing of KLN-1010
  All adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) or American Society for Transplantation and Cell Therapy (ASTCT) criteria

SECONDARY OUTCOMES:
Pharmacokinetics of KLN-1010 after dosing. | Up to two years after dosing with study drug.
  Peak of virus vector genomes (Cmax of lentivirus) in blood.
Pharmacokinetics of KLN-1010 (Tmax). | Up to two years after infusion with study drug.
  Measurement of time to the highest amount of viral vector in the blood.
Pharmacokinetics of KLN-1010 Area Under the Curve (AUC) | Up to two years after infusion with study drug.
  Measurement of the amount of viral vector (AUC of lentivirus) in blood over time.
Pharmacokinetics of CAR-T cells generated. | Up to two years after infusion with study drug.
  The presence and number of CAR-T (Cmax) cells present in blood.
Pharmacokinetics of CAR-T cells generated (Tmax). | Up to two years after infusion with study drug.
  Measurement of time to the highest amount of CAR-T cells in the blood.
Pharmacokinetics of CAR-T cells generated Area Under the Curve (AUC) | Up to two years after infusion with study drug.
  Measurement of the amount of CAR-T cell DNA in blood and bone marrow over time.
Assessment of Multiple Myeloma | From dosing until disease progression or up to 15 years from receiving study drug, whichever happens first.
  Participants will have multiple myeloma assessed according to the International Myeloma Working Group (IMWG) response criteria.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - The Royal Prince Alfred, Camperdown, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Paula Fox Melanoma and Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Kelonia will make individual anonymized participant data available to qualified researchers.